CLINICAL TRIAL: NCT04540055
Title: Effects of General Anesthesia vs. General Anesthesia and Paravertebral Block to IL-2, IL-6, PGE2, MMP-9, and Clinical Outcome in Modified Radical Mastectomy
Brief Title: General Anesthesia and Paravertebral Blocks vs. General Anesthesia Only: Influence Inflammation Factors and Clinical Outcomes in Modified Radical Mastectomy
Status: Completed | Type: Observational
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Christopher Ryalino, Lecturer, Udayana University
Other Study IDs: UNUD-CTR-FK300820-004
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Anesthesia, Local; Anesthesia; Inflammatory Response; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paravertebral (Group P): Patients underwent MRM under the combination of general anesthesia and paravertebral block.
  Interventions: Procedure: Paravertebral block
- General Anesthesia (Group G): Patients underwent MRM under general anesthesia.
  Interventions: Procedure: General Anesthesia

INTERVENTIONS:
Procedure: Paravertebral block — The subjects in this group received general anesthesia and USG-guided paravertebral block
  Groups: Paravertebral (Group P)
Procedure: General Anesthesia — The subjects in this group underwent MRM under routine general anesthesia without peripheral nerve block supplementation.
  Groups: General Anesthesia (Group G)

SUMMARY:
Regional anesthesia and analgesia may maintain immune function, reduce surgical stress, and also reduce volatile anesthetics and opioids requirements. Local anesthetic drugs used in regional anesthesia and analgesia work to have anti-proliferative and cytotoxic effects on cancer cells. Pro-inflammatory cytokines such as IL-1, IL-6, and TNF-alpha increase in levels in peripheral nerves, spinal cord, brain (brain stem, locus sereleus, thalamus, hippocampus, and prefrontal cortex) after peripheral nerves are injured. The anti-inflammatory cytokine IL-10 is decreased in levels after peripheral nerve injury. The balance between pro-inflammatory and anti-inflammatory cytokines affects the severity of pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient with breast cancer (stadium Ia, Ib, IIa, IIb, IIIa, IIIb) undergoing MRM surgery
* Balinese race
* ASA physical status I, II, III

Exclusion Criteria:

* History of allergy to drugs used in anesthesia
* History psychiatric disorder
* History of perioperative transfusion
* History of autoimmune disease
* History of taking beta blockers or anti-platelet aggregation medications
* Previous breast surgery
* Spine deformity
* Coagulopathy
* Local infections in paravertebral block site
* Decreased renal function
* Neurological deficits
* Peptic ulcer

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer (stadium Ia-IIIb) who underwent MRM surgery under general anesthesia in Sanglah General Hospital
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Concentration of IL-2 in blood serum | 1-hour after surgery
  Concentration of IL-2 level in blood serum
Concentration of IL-2 in blood serum | 24-hours after surgery
  Concentration of IL-2 level in blood serum
Concentration of IL-6 in blood serum | 1-hour after surgery
  Concentration of IL-6 level in blood serum
Concentration of IL-6 in blood serum | 24-hours after surgery
  Concentration of IL-6 level in blood serum
Visual Analog Scale (VAS) | 24-hours after surgery
  pain score measured by visual analog scale (VAS), scaled between 0 (no pain) and 10 (worst pain)

SECONDARY OUTCOMES:
Concentration of PGE2 level in blood serum | 1-hour after surgery
  Concentration of PGE2 level in blood serum
Concentration of PGE2 level in blood serum | 24-hours after surgery
  Concentration of PGE2 level in blood serum
Concentration of MMP-9 level in blood serum | 1-hour after surgery
  Concentration of MMP-9 level in blood serum
Concentration of MMP-9 level in blood serum | 24-hours after surgery
  Concentration of MMP-9 level in blood serum

CONTACTS AND LOCATIONS:
Locations (1):
- Sanglah General Hospital, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided